CLINICAL TRIAL: NCT05046990
Title: Arrangement of Collecting Venules for the Endoscopic Diagnosis of Helicobacter Pylori Infection (MOTIVATION): International Multicentre Study Outside Asia
Brief Title: Arrangement of Collecting Venules for the Endoscopic Diagnosis of Helicobacter Pylori
Acronym: MOTIVATION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: HCB-RAC-MOTIVATION
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-12

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RAC evaluation: Patients older than 18 years without previous history of Hp infection or eradication undergoing a gastroscopy
  Interventions: Diagnostic Test: Regular Arrangement of Collecting Venules

INTERVENTIONS:
Diagnostic Test: Regular Arrangement of Collecting Venules — This is a prospective, multicentre, international study without a control group.

SUMMARY:
To perform a prospective, observational, international, multicentre, in vivo study to assess the performance of regular arrangement of collecting venules (RAC) for the exclusion of Helicobacter pylori (Hp) infection using white light high definition (HD) endoscopy without any kind of zoom or magnification.

Gold standard will be mucosal biopsies (Sydney protocol) or urease test. Immunohistochemistry (IHC) should be performed in case of a negative histologic study for Hp in patients taking proton pump inhibitors (PPIs).

Participants will perform a training test with 20 pictures of the distal part of the lesser curvature before starting the inclusion of cases.

Secondary objectives are:

* To assess whether age, sex and PPIs, have an influence on the results of RAC.
* To assess the correlation of atrophic gastritis and intestinal metaplasia (confirmed in histopathological samples) and RAC.
* To assess reproducibility of RAC on real time examinations with different operators and in different countries with different Hp infection prevalence.

Primary and secondary variables

The primary study variable is:

- Endoscopic detection of RAC.

Secondary variables will be considered:

* Sex
* Age
* PPI intake in the last two weeks
* Centre
* Country
* Hp prevalence
* Endoscopist
* Type of endoscope
* Significant findings (need of histological confirmation)

  * Atrophic gastritis
  * Intestinal metaplasia
  * Erosive gastritis
  * Benign gastric ulcer
  * Gastric adenoma
  * Gastric cancer

DETAILED DESCRIPTION:
This is a prospective, multicentre, international study without a control group.

Training phase Before starting the inclusion of patients, 20 HD images previously collected by the principal investigator will be sent to each of the study investigators. Pictures will clearly show the RAC pattern present or absent at the level of the distal gastric lesser curvature. In case of doubtful RAC, the pattern shall be considered negative. Investigators will be able to discuss their questions and doubts after the training phase (videoconference).

Endoscopic examination Upper endoscopy will be performed with HD endoscopes and a high-definition screen. Two endoscopists will participate in each hospital. The examination will be performed according to the protocol of each centre. Visualisation of the entire oesophageal, gastric and duodenal surface will be performed as in routine clinical practice. The presence of RAC will be assessed during the gastric exploration with sufficient insufflation and its detection will be considered as the presence of a regular starfish-shaped erythematous punctation in the lower part of the lesser curvature of the gastric body, close to the incisura angularis.

In case of the presence of residues in the gastric cavity that prevent the correct visualisation of the area, water washings shall be performed for the correct characterisation of the mucosa. At least one photo of the described gastric region shall be taken with the image processor system to maintain its high-definition quality. All the data (name, date of birth, clinical record number, date of exploration…) will be removed from the picture to ensure the anonymisation. Subsequently, the photographs will be downloaded and saved in a folder on a network drive of each hospital.

After characterisation of the gastric mucosa, the Hp infection status will be assessed by taking biopsies with a standard forceps for anatomopathological study according to Sydney's protocol (2 in the antrum, 1 in the incisura and 2 in the body). Ideally, biopsies for a urease test will also be obtained.

Histopathological examination Samples shall be fixed in formalin and analysed by the Anatomical Pathology service for histological examination by haematoxylin and eosin (H&E) and special staining for Hp (e.g. modified Giemsa). In patients taking PPI, if Hp is negative in the H&E histological study, the study will be completed by immunohistochemical (IHC) staining.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years without previous history of Hp infection or eradication undergoing a gastroscopy

Exclusion Criteria:

* Patients taking oral anticoagulants (acenocoumarol and new anticoagulants as dabigatran, rivaroxaban, apixaban and edoxaban), NSAIDs or with intake of antibiotics in the last 4 weeks, but aspirin at a dose of 100 mg per day will be included
* Diseases that affect the gastric mucosa and preclude the evaluation of the collecting venules pattern (portal hypertension, gastric lymphoma)
* History of previous gastric cancer or patients in surveillance for preneoplastic lesions (atrophic gastritis/IM),
* Previous gastric surgery,
* Active bleeding or presence of blood or food that would impede a complete mucosal evaluation.
* Negative to participate in the study or inability to provide signed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years without previous history of Hp infection or eradication undergoing a gastroscopy in each center
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
RAC performance | 12 months
  A total of 1000 consecutive patients with no history of Hp who come for gastroscopy will be included in the study to perform a prospective, observational, international, multicentre, in vivo study to assess the performance of regular arrangement of collecting venules (RAC).
  Endoscopists will perform a training test with 20 pictures of the distal part of the lesser curvature before starting the inclusion of cases. 17 different centers will participate in the study and each of them will include between 50 and 100 patients.
  Presence of RAC using white light high definition endoscopy without magnification determines the exclusion of Helicobacter pylori (Hp) infection. Gold standard diagnosis test for Hp infection will be histological results by mucosal biopsies (Sydney protocol) or urease test. Immunohistochemistry (IHC) should be performed in case of a negative histologic study for Hp in patients taking proton pump inhibitors (PPIs).

SECONDARY OUTCOMES:
Baseline characteristics | 12 months
  To assess whether age, sex and PPIs, have an influence on the results of RAC in all patients.
Histological correlation | 12 months
  To assess the correlation of atrophic gastritis and intestinal metaplasia (confirmed in histopathological samples) and RAC in all patients.
Reproducibility | 12 months
  To assess reproducibility of RAC on real time examinations with different operators and in different countries with different Hp infection prevalence.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Fernandez-Esparrach, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (5):
- Cliniques Universitaires Saint Luc, Brussels, Belgium
- München University Hospital, Munich, Bavaria, Germany
- Spain (3):
  - Hospital de Mérida, Mérida, Badajoz
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital Clinic de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garces-Duran R, Galdin-Ferreyra M, Delgado-Guillena PG, Cuatrecasas M, Cordova H, Garcia-Rodriguez A, Rodrigo-Calvo MT, Jimeno-Ramiro M, Araujo IK, Gines A, Llach J, Fernandez-Esparrach G. Diagnosis of Helicobacter pylori Infection by the Arrangement of Collecting Venules Using White Light Endoscopy: Evaluation of Interobserver Agreement. Dig Dis. 2022;40(3):376-384. doi: 10.1159/000518100. Epub 2021 Jun 30. PMID 34348294
- [Background] Garces-Duran R, Garcia-Rodriguez A, Cordova H, Cuatrecasas M, Gines A, Gonzalez-Suarez B, Araujo I, Llach J, Fernandez-Esparrach G. Association between a regular arrangement of collecting venules and absence of Helicobacter pylori infection in a European population. Gastrointest Endosc. 2019 Sep;90(3):461-466. doi: 10.1016/j.gie.2019.05.027. Epub 2019 May 17. PMID 31108089